CLINICAL TRIAL: NCT03255005
Title: A Controlled Study to Evaluate the Efficacy of an Endoluminal-suturing Device (Endomina) as an Aid for Endoscopic Gastric Reduction
Brief Title: Endomina Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P2017/401
Record Dates: First submitted 2017-08-08; First posted 2017-08-21 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Obesity
Keywords: obesity; endoscopy; endoscopic sleeve gastroplasty
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Group A: treatment J0 + Diet 1 year Group B: Diet 6 months - Treatment - Diet 1 year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Endoscopic sleeve gastroplasty (Endomina) at J0 with multidisciplinary follow-up for 1 year
  Interventions: Device: Endomina
- Controled group (Active Comparator): Diet for 6 months then Endoscopic sleeve gastroplasty (Endomina) with multidisciplinary follow-up for 1 year
  Interventions: Device: Endomina; Behavioral: Diet

INTERVENTIONS:
Device: Endomina — Endoscopic sleeve reduction
Behavioral: Diet — Multidisciplinary follow-up
  Arms: Controled group

SUMMARY:
The aim of this trial is to evaluate the efficacy of an endoluminal vertical gastroplasty (EVG) using an endoluminal-suturing device. Safety will also be characterized, in particular by the incidence of all Adverse Device Effects (ADEs). A secondary endpoint is to compare a delayed treatment control group (diet alone; crossover at 6 months) with a treatment group (EVG plus diet). Other secondary endpoints include improvements in other obesity measures.

DETAILED DESCRIPTION:
Surgery is currently the only effective treatment for morbid obesity and can be divided into restrictive surgeries (Lap Band and Sleeve gastrectomy), malabsorptive surgeries (Biliary pancreatic deviation and duodenal switch) or a combination of both (RYGBP).

This latter technique is the most common and most effective surgical procedure performed worldwide and has been processed to be an effective treatment of morbid obesity and its complications, achieving excess weight loss of 65 to 80 %; 1-2 years after surgery.

Vertical gastric plication is a novel surgical approach for reducing the stomach capacity. Anterior surface plication and greater curvature plication are variations of vertical gastric plication that reduce the gastric capacity through infolding of the anterior surface or greater curvature of the stomach, respectively. These approaches have been tested, with positive results.

A transoral or endoluminal approach (i.e. a procedure that requires no incision, because access is granted through the mouth) offers the potential for additional benefit to the patient, because the procedures continue to become more and more minimally invasive.

Advances in endoluminal devices are now allowing clinicians the ability to begin exploring bariatric procedures performed via flexible endoscopy. Although these procedures may not be as effective as their surgical counterparts, these less-invasive options may relieve patients of the significant risks associated with surgery and might become part of the armamentarium of obesity management.

Endomina (Endo Tools Therapeutics, Gosselies, Belgium) is a CE marked device that may be attached to an endoscope inside the body and allows remote actuation of the device during a peroral intervention. It offers the possibilities of making transoral full thickness tissue apposition and may allow performing, via a transoral route, large plications with tight serosa to serosa apposition.

After a first trial on pigs (safety), a second trial on human patients was performed. This trial included 11 patients treated with the same technique. There were no complications and the short term results were encouraging with 41% EWL at 6 month.

A multicentric trial NCT02582229 entitled: " A Prospective Study to Evaluate the Efficacy of an Endoluminal-suturing Device (Endomina TM) as an Aid for Endoscopic Gastric Reduction. " is ongoing and inclusion of patients ended in December 2016 with a total of 51 patients included in 3 European centers. Early results of the trial had showed that dietician follow-up is an important part of the success. During that time implementation of the procedure had been done.

The aim of this trial is to compare a control group (diet alone) with a treatment group (Endomina procedure plus diet).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years;
2. Class I or class II obesity (i.e. BMI between 30 to 40 kg/m²);
3. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment, endoscopy, radiography, as well as laboratory investigations;
4. Must be able to understand and be willing to provide written informed consent;
5. Must live within 75 km of the treatment site;
6. Had followed the bariatric multidisciplinary workup (blood analyses, dietician, psychologist and doctor appointments).

Exclusion Criteria:

1. Achalasia and any other esophageal motility disorders;
2. Severe esophagitis;
3. Gastro-duodenal ulcer;
4. Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity;
5. Hypertension: uncontrolled hypertension during last 3 months;
6. Diabetes: uncontrolled diabetes (on insulin therapy or oral therapy with Hba1c > 10%);
7. TBWL >5% over the last 6 months;
8. Severe renal, hepatic, pulmonary disease or cancer;
9. GI stenosis or obstruction;
10. Pregnancy, breastfeeding or willing to become pregnant in the coming 18 months;
11. Previous bariatric surgery, balloon or other endoscopic obesity-related therapy;
12. Anticoagulant therapy;
13. Impending gastric surgery 60 days post intervention;
14. Currently participating in other study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of all Adverse Device Effects | one year from procedure
  Safety will be characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants.
Weight loss | one year from procedure
  total weight loss and excess weight loss

SECONDARY OUTCOMES:
Weight loss at 6 months | at 6 months after the procedure (treatment group)
  comparison between diet and treatment group at 6 months
More than 15% weight loss | one year from procedure
  Proportion of patients in the Endomina Group with a loss of weight of more than 15%
Quality of life | one year from procedure
  SF36
TBWL | one year from procedure
  Mean % total body weight loss (%TBWL)
Weight and height | one year from procedure
  To calculate the body mass index (BMI)

CONTACTS AND LOCATIONS:
Locations (2):
- Gastroenterology Department Erasme Hospital, Brussels, Belgium
- APHM Hopital Marseille Nord Hepato-Gastroentérologie et Oncologie Digestive, Marseille, France

REFERENCES:
- [Result] ASGE Bariatric Endoscopy Task Force and ASGE Technology Committee; Abu Dayyeh BK, Kumar N, Edmundowicz SA, Jonnalagadda S, Larsen M, Sullivan S, Thompson CC, Banerjee S. ASGE Bariatric Endoscopy Task Force systematic review and meta-analysis assessing the ASGE PIVI thresholds for adopting endoscopic bariatric therapies. Gastrointest Endosc. 2015 Sep;82(3):425-38.e5. doi: 10.1016/j.gie.2015.03.1964. Epub 2015 Jul 29. PMID 26232362
- [Result] Magro DO, Geloneze B, Delfini R, Pareja BC, Callejas F, Pareja JC. Long-term weight regain after gastric bypass: a 5-year prospective study. Obes Surg. 2008 Jun;18(6):648-51. doi: 10.1007/s11695-007-9265-1. Epub 2008 Apr 8. PMID 18392907
- [Result] Menchaca HJ, Harris JL, Thompson SE, Mootoo M, Michalek VN, Buchwald H. Gastric plication: preclinical study of durability of serosa-to-serosa apposition. Surg Obes Relat Dis. 2011 Jan-Feb;7(1):8-14. doi: 10.1016/j.soard.2010.11.002. Epub 2010 Nov 12. PMID 21255733
- [Result] Fogel R, De Fogel J, Bonilla Y, De La Fuente R. Clinical experience of transoral suturing for an endoluminal vertical gastroplasty: 1-year follow-up in 64 patients. Gastrointest Endosc. 2008 Jul;68(1):51-8. doi: 10.1016/j.gie.2007.10.061. Epub 2008 Mar 19. PMID 18355825
- [Result] Paxton JH, Matthews JB. The cost effectiveness of laparoscopic versus open gastric bypass surgery. Obes Surg. 2005 Jan;15(1):24-34. doi: 10.1381/0960892052993477. PMID 15760496
- [Result] Huberty V, Ibrahim M, Hiernaux M, Chau A, Dugardeyn S, Deviere J. Safety and feasibility of an endoluminal-suturing device for endoscopic gastric reduction (with video). Gastrointest Endosc. 2017 Apr;85(4):833-837. doi: 10.1016/j.gie.2016.08.007. Epub 2016 Aug 22. PMID 27562938
- [Result] ASGE Bariatric Endoscopy Task Force; ASGE Technology Committee; Abu Dayyeh BK, Edmundowicz SA, Jonnalagadda S, Kumar N, Larsen M, Sullivan S, Thompson CC, Banerjee S. Endoscopic bariatric therapies. Gastrointest Endosc. 2015 May;81(5):1073-86. doi: 10.1016/j.gie.2015.02.023. Epub 2015 Mar 28. No abstract available. PMID 25828245
- [Result] ASGE/ASMBS Task Force on Endoscopic Bariatric Therapy; Ginsberg GG, Chand B, Cote GA, Dallal RM, Edmundowicz SA, Nguyen NT, Pryor A, Thompson CC. A pathway to endoscopic bariatric therapies. Gastrointest Endosc. 2011 Nov;74(5):943-53. doi: 10.1016/j.gie.2011.08.053. No abstract available. PMID 22032311
- [Result] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Derived] Huberty V, Boskoski I, Bove V, Van Ouytsel P, Costamagna G, Barthet MA, Deviere J. Endoscopic sutured gastroplasty in addition to lifestyle modification: short-term efficacy in a controlled randomised trial. Gut. 2020 Oct 28:gutjnl-2020-322026. doi: 10.1136/gutjnl-2020-322026. Online ahead of print. PMID 33115727